CLINICAL TRIAL: NCT00976261
Title: A 2-Part Trial: a Randomized 6-day Repeat-dose, Parallel-group Study in Subjects With T2DM to Assess the Safety and Tolerability of GSK1614235 Compared to Placebo and Sitagliptin; and a Randomized Single-dose, Food Effect Study in Healthy Volunteers to Assess Safety and Tolerability of GSK1614235
Brief Title: A 2-Part Trial in Subjects With Type 2 Diabetes and in Healthy Subjects to Evaluate GSK1614235, a New Glucose Lowering Drug to Treat Type 2 Diabetes
Acronym: SGA112534
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 112534
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; single dose; 3-O-methylglucose; healthy volunteer; repeat dose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK1614235 (Experimental): Glucose lowering agent under investigation.
  Interventions: Drug: GSK1614235
- Sitagliptin (Active Comparator): Glucose lowering comparator
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo to match GSK1614235 and placebo to match Sitagliptin
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GSK1614235 — Glucose lowering in Type 2 Diabetes Mellitus
  Other Names: Type 2 Diabetes Mellitus
  Arms: GSK1614235
Drug: Sitagliptin — Glucose lowering in Type 2 Diabetes Mellitus
  Other Names: Type 2 Diabetes Mellitus
  Arms: Sitagliptin
Other: Placebo — Comparator
  Other Names: Type 2 Diabetes Mellitus
  Arms: Placebo

SUMMARY:
The purpose of Part A of this study is to test whether repeated doses of the study drug (GSK1614235) are safe and well tolerated (i.e. do not produce unacceptable side effects) and whether we can obtain some preliminary information as to whether it works in lowering blood glucose levels. We will do this by comparing the effect of the study drug with placebo (no drug present) and against a drug (sitagliptin) known to control blood glucose in the treatment of diabetes.

The purpose of Part B of this study is to determine the how the timing of dosing, relative to meals, affects the response to study drug.

DETAILED DESCRIPTION:
Part A is a double-blind, randomized, parallel group, dose-ranging study, in subjects with type 2 diabetes mellitus to assess safety, tolerability, and to estimate the pharmacodynamic effects when subjects receive repeated doses of placebo, sitagliptin (Januvia), or GSK1614235. The target is to explore the best doses of GSK1614235 that provide glucose control with minimal adverse effects.

There will be at least 4 cohorts of subjects:

* Cohort 1: 8 subjects randomized to receive placebo, 100mg sitagliptin QD, or 1mg GSK1612435 BID
* Cohort 2: 6 subjects randomized to receive placebo, 100mg sitagliptin QD, or 5mg GSK1612435 BID.
* Cohort 3: 6 subjects randomized to receive placebo, 100mg sitagliptin QD, or 20mg GSK1612435 BID.
* Cohort 4: 20-40 subjects randomized to receive placebo, 100mg sitagliptin QD, or GSK1612435 BID, (potential doses of 0.25 to 40mg BID), depending on safety, tolerability, and glucose results of Cohorts 1, 2, and 3.
* Cohort 5: 12 subjects randomized to receive placebo or GSK1614235 BID (potential doses of up to 80mg BID), depending on safety, tolerability, and glucose results of Cohorts 1, 2, 3, and 4.
* Cohort 6: 24 subjects randomized to receive GSK1614235 BID (20BID), or sitagliptin (100mg QD).

After subjects have successfully completed the screening procedures, they will be asked to discontinue prior anti-diabetic therapy at least 72 h before admission to the research facility and remain off of the medications until the completion of the follow-up visit (total of ~14 days). Subjects will be admitted to the research facility on the evening of Day -2 in preparation to begin baseline assessments, including PD, on Day -1 (for their particular cohort). Beginning on Day 1, subjects will receive a single dose of GSK1614235 and undergo PK sampling, and on Day 2 through Day 6, subjects will be dosed on a twice daily dosing schedule with doses administered immediately before breakfast and the evening meal. Day 6 includes intensive assessments of PK and PD parameters in addition to routine safety monitoring.

Part B is a double-blind, randomized, single-dose, 3-way crossover study in 12 subjects. A well-tolerated dose of GSK1614235 that provides a meaningful pharmacodynamic response based on data from Part A will be administered in both fed and fasted states. It is not anticipated that the dose for Part B will exceed single doses of 40mg.

Part B will consist of 3 periods. Period 1 will begin after subjects have successfully completed screening. They will be admitted to the research facility the evening before dosing (Day -1) and will dose the following morning after an overnight (at least 12 hour fast). Safety monitoring and PK and PD sampling will be conducted over a 48 hour period. Subjects will be discharged from the research facility after the 48 hour PK and PD sample has been collected. A washout period of ≥ 5 days period will ensue, and subjects will be admitted to the research facility to begin Period 2. Period 3 will follow the same schedule as Period 1 and Period 2.

Subjects will be randomized such that, at separate admissions, each subject receives the selected GSK1614235 dose or matching placebo as follows.

* GSK1614235 before meal and placebo after meal
* GSK1614235 30 min after meal and placebo before meal
* Placebo - both before meal and 30 min after meal

ELIGIBILITY:
Inclusion Criteria Part A:

* Subjects with documented type 2 diabetes mellitus diagnosis whose HbA1c levels are >7 and at or less than 9.5%; at screening, who are either controlled by diet alone, or are on monotherapy with oral sulfonylureas, DPP-IV inhibitors (e.g. sitagliptin), or metformin.
* Men and women 30 - 65 years of age, inclusive, at screening.
* Women: post-menopausal or surgically sterile, i.e. women of non-childbearing potential.
* Male subjects must agree to use a contraception method
* Body weight 50kg for men and 45kg for women and BMI within the range 22 35kg/m2, inclusive.
* Subjects taking stable regimens of aspirin, ACE inhibitors, beta-blockers, calcium channel blockers, thyroid replacement hormone, and HMG-CoA reductase inhibitors (statins) will be allowed if their dose regimen(s) remain constant throughout the study period.
* Signed and dated written informed consent prior to enrollment into the study, including performance of any screening procedures.
* The subject is able to understand and comply with protocol requirements
* In France, a subject will be eligible for inclusion in this study if he or she is affiliated with or a beneficiary of a social security category.

Exclusion Criteria Part A:

* Requiring insulin therapy or use of combination oral antidiabetic medications or use of monotherapy other than oral sulfonylureas, DPP-IV inhibitors (e.g. sitagliptin), or metformin within the 3 months prior to screening.
* Medically unable or unwilling to discontinue current anti-diabetic therapy for 72 hours prior to admission to the research facility and remain off medication until the follow-up visit.
* Past or present disease (other than type 2 diabetes mellitus) including, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease and endocrine disease.
* Past or present history of irritable bowel syndrome, gastrointestinal surgeries, or any other gastrointestinal complaints, history of GI intolerance to sitagliptin, lactose intolerance or hepatobiliary conditions that may interfere with the absorption of GSK1614235 or interfere with the objectives and endpoints of the study.
* As a result of the medical interview and/or the physical examination, Investigator considers the subject inappropriate for inclusion in the study.
* History or presence of sensitivity or allergy to the study drug or drugs, GSK 1614235 or sitagliptin, their components, or drugs of these classes or a history of drug or other allergy that contraindicates participation.
* Subjects with laboratory results that are not clinically significant may be included in the study
* Significant renal disease as manifested by one of the following:

Creatinine clearance <60mL/min Urine albumin concentration at or >300ug/mg of creatinine. Known loss of a kidney, either by surgical ablation, injury, or disease.

* Positive test results for hepatitis C antibodies, hepatitis B surface antigen, and HIV at screening.
* Abuse of alcohol
* A positive pre-study urine drug screen
* No significant concomitant health problems other than type 2 diabetes mellitus and otherwise healthy. Subjects with the following clinical laboratory values are excluded:

ALT or AST > 2 times the upper limit of normal at screening. Bilirubin > 1.5 times the upper limit of normal at screening (total; subjects above this limit may only be included if direct bilirubin is within normal limits).

Fasting triglycerides > 400mg/dL (22.2mmol/L) at screening. Fasting LDL cholesterol > 160mg/dL (3.3mmol/L). Participation in a study trial with any investigational new drug (new chemical entity) within 90 days prior to the start of the study.

For ECG rates and intervals, the average of 3 ECG assessments, separated by 5 minutes is used. Significant ECG abnormalities include but are not limited to:

Males Females Heart Rate < 45 and >100 bpm < 45 and >100 bpm PR Interval <120 and > 220 ms <120 and > 220 ms QRS duration < 70 and >120 ms < 70 and >120 ms QTC Interval (Bazett) > 450 ms > 450 ms

* Blood pressure must be at or >80/60mmHg and at or <150/95mmHg at screening and at admission to the study facility.
* Participation in the study will result in the subject having donated more than 1,500mL blood (males) or 1,000mL (females) in the previous 12 months and where participation in study would result in donation of blood in excess of 580mL within a 56-day period.
* Participation in a study trial with any investigational new drug (new chemical entity) within 90 days prior to the start of the study.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless it is in the opinion of the investigator and sponsor that the medication will not interfere with 17. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* otinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Inclusion Criteria Part B:

* Healthy as determined by medical evaluation: medical history, physical examination, ECG, and laboratory tests. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the finding is unlikely to introduce additional risk and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Body weight at or >50 kg for men, at or >45kg for women, and BMI within the range 19 - 30 kg/m2 (inclusive).
* A female subject is eligible to participate if she is of non-childbearing potential
* Male subjects must agree to use a contraception method
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Part B Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Past or present disease that may affect the outcome of this study, including, but not limited to: cardiovascular, renal, hepatic, malignancy, hematological, neurological, and/or endocrine.

Clinically significant abnormalities are noted for ECG assessments. For rates and intervals, the average of 3 ECG assessments, separated by 5 minutes is used. Significant ECG abnormalities include but are not limited to:

Males Females Heart Rate < 45 and >100 bpm < 45 and >100 bpm PR Interval <120 and > 220 ms <120 and > 220 ms QRS duration < 70 and >120 ms < 70 and >120 ms QTC Interval (Bazett) > 450 ms > 450 ms

* Past or present history of irritable bowel syndrome, gastrointestinal surgeries, or any other gastrointestinal complaints, history of GI intolerance to sitaglitpin, lactose intolerance or hepatobiliary conditions that may interfere with the absorption of GSK1614235 or interfere with the objectives and endpoints of the study.
* AST, ALT, alkaline phosphatase or bilirubin > 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Fasting triglycerides > 400mg/dL at screening
* Fasting LDL cholesterol > 160mg/dL
* Clinically significant abnormalities of TSH or known thyroid disease.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Participation in a clinical trial and received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that contraindicates participation.
* Participation in the study will result in the subject having donated more than 1,500mL blood (males) or 1,000mL (females) in the previous 12 months and where participation in study would result in donation of blood in excess of 580mL within a 56-day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-10-17 (Actual); Primary Completion 2010-09-05 (Actual); Study Completion 2010-09-05 (Actual)

PRIMARY OUTCOMES:
Part A: Safety, tolerability parameters: adverse events, gastro-intestinal side effects, subject reported outcomes, clinical laboratory results, ECGs and vital signs | 6 days
Part B: Safety, tolerability parameters: adverse events, gastro-intestinal side effects, subject reported outcomes, clinical laboratory results, ECGs and vital signs | 1 day

SECONDARY OUTCOMES:
Part A: Pharmacokinetics | 6 days
Part A: Pharmacodynamics | 6 days
Part B: Pharmacokinetics | 1 day
Part B: Pharmacodynamics | 1 day
Part B: 3-O-Methyl-Glucose Kinetics | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (3):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Cincinnati, Ohio
- France (2):
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Rueil-Malmaison
- Germany (3):
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Dobbins RL, Greenway FL, Chen L, Liu Y, Breed SL, Andrews SM, Wald JA, Walker A, Smith CD. Selective sodium-dependent glucose transporter 1 inhibitors block glucose absorption and impair glucose-dependent insulinotropic peptide release. Am J Physiol Gastrointest Liver Physiol. 2015 Jun 1;308(11):G946-54. doi: 10.1152/ajpgi.00286.2014. Epub 2015 Mar 12. PMID 25767259
- See also: Results for study 112534 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/112534?search=study&study_ids=112534#rs